CLINICAL TRIAL: NCT06681155
Title: A Prospective Cohort Study on the Identification of High-Risk Coronary Plaque by Multimodality Intravascular Imaging(PlaqueVision Study)
Brief Title: Identification Of High-risk Coronary Plaques By Multimodal Intravascular Imaging
Acronym: PlaqueVision
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yun Dai Chen, Principal Investigator, Chinese PLA General Hospital
Other Study IDs: HZKY-PJ-2024-54
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Coronary Arterial Disease (CAD); Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-risk Plaque Group: Multimodal intravascular imaging technology is used to assess the morphological structure and stability of non-criminal lesions in plaques, categorized into high-risk and non-high-risk groups. High-risk plaques are defined as those that meet any of the following criteria: ① IVUS minimum lumen area <4.0mm² or OCT minimum lumen area <3.5mm², ② plaque burden >70%, ③ presence of thin-cap fibroatheroma, ④ NIRS detects lipid-rich plaques with LRP MaxLCBI4mm >315, and are considered high-risk if they have at least two of the above four characteristics. A patient is placed in the high-risk group if they have at least one high-risk plaque.
  Interventions: Diagnostic Test: Assessment of plaque morphology, structure, and stability in non-culprit lesions
- Non-high-risk Plaque Group: Multimodal intravascular imaging technology is used to assess the morphological structure and stability of non-criminal lesions in plaques, categorized into high-risk and non-high-risk groups. High-risk plaques are defined as those that meet any of the following criteria: ① IVUS minimum lumen area <4.0mm² or OCT minimum lumen area <3.5mm², ② plaque burden >70%, ③ presence of thin-cap fibroatheroma, ④ NIRS detects lipid-rich plaques with LRP MaxLCBI4mm >315, and are considered high-risk if they have at least two of the above four characteristics. If they have no high-risk plaques, they are placed in the non-high-risk group.
  Interventions: Diagnostic Test: Assessment of plaque morphology, structure, and stability in non-culprit lesions

INTERVENTIONS:
Diagnostic Test: Assessment of plaque morphology, structure, and stability in non-culprit lesions — Assessment of plaque morphology, structure, and stability in non-culprit lesions based on intravascular ultrasound and optical coherence tomography-near-infrared spectroscopy imaging technology.

SUMMARY:
This study is a multicenter prospective observational clinical study, which will be conducted in 11 hospitals, and approximately 500 subjects will be enrolled. Plaque morphology and stability of non-culprit lesions were assessed by intravascular ultrasound (IVUS) and optical coherence tomography-near-infrared spectroscopy (OCT) after percutaneous coronary intervention (PCI) in patients with acute coronary syndrome (ACS). Plaques were grouped according to high-risk or non-high-risk. Clinical follow-up was conducted after PCI.

DETAILED DESCRIPTION:
Plaque stability is an important criterion for selecting different treatment strategies (interventional and antithrombotic). High-risk plaque characteristics are also considered to be related to the overall incidence of Major Adverse Cardiovascular Events (MACE). Single-modality intravascular imaging has inherent disadvantages in identifying atherosclerotic plaques, while the combination of IVUS, OCT, and NIRS enables multimodal intravascular imaging techniques to complement each other in obtaining plaque information. There is currently a lack of research on the prognostic benefits of multimodal intravascular imaging in assessing atherosclerotic plaques. This study is a multicenter, prospective, observational clinical study that will be conducted at 11 hospitals, enrolling approximately 500 subjects. It will use intravascular ultrasound (IVUS) and optical coherence tomography-near-infrared spectroscopy (OCT) to assess the morphology and stability of non-culprit lesions in patients with acute coronary syndrome (ACS) after percutaneous coronary intervention (PCI), and will follow up at 1 month, 1 year, 2 years, and 5 years post-surgery. The aim is to compare the clinical outcomes between high-risk and non-high-risk patients, as well as between high-risk and non-high-risk plaques defined by multimodal intravascular imaging, and to explore the predictive value of high-risk plaque characteristics shown by multimodal intravascular imaging for adverse cardiovascular events in patients with ACS.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the clinical study:

  1. Aged ≥18 years at enrollment, male or female;
  2. Meets the diagnosis of acute coronary syndrome, including acute myocardial infarction and unstable angina. Acute myocardial infarction includes ST-elevation myocardial infarction (STEMI) and non-ST-elevation myocardial infarction (non-STEMI). STEMI is defined as chest pain lasting at least 30 minutes, arriving at the hospital within 12 hours from the onset of symptoms, changes in the 12-lead ECG (ST-segment elevation >0.1 mV in ≥2 consecutive leads or new left bundle branch block), and elevated cardiac biomarkers (troponin T/I). Non-STEMI is defined as ischemic symptoms without ST-segment elevation on ECG, accompanied by elevated cardiac biomarkers. Unstable angina is defined as chest pain lasting 5-30 minutes at rest, or worsening of exertional angina, and accompanied by one of the following: transient ST-segment depression or elevation; coronary angiography showing luminal narrowing ≥90% or plaque rupture or thrombotic lesions.
  3. Planned to undergo coronary angiography and PCI treatment;
  4. Hemodynamically stable and able to tolerate repeated intracoronary administration of nitroglycerin;
  5. Capable of understanding the requirements of this study, willing to participate in the study, and have signed an informed consent form.
* Imaging inclusion criteria:

  1. Coronary angiography clearly shows that the patient has at least one non-culprit lesion with a visual assessment of diameter stenosis between 40-70%, and the operator believes that interventional treatment intervention is not temporarily necessary;
  2. The site of the non-culprit lesion has not previously had a stent implanted.

Exclusion Criteria:

* Exclusion criteria for the clinical study:

  1. Cardiogenic shock or hemodynamic instability;
  2. History of coronary artery bypass grafting (CABG), or planned CABG;
  3. Severe renal impairment (glomerular filtration rate <30ml/min/1.73m²);
  4. Life expectancy of less than 2 years;
  5. Currently participating in other ongoing investigative device or drug studies that have not yet reached their primary endpoints.
* Imaging exclusion criteria:

The anatomical structure of the non-culprit lesion is not suitable for intravascular imaging catheter imaging (lesions at the left main trunk or right coronary artery ostium, severe calcification, chronic total occlusion, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Coronary Syndrome (ACS) who are planned for coronary angiography and interventional treatment. ACS includes acute ST-segment elevation myocardial infarction, acute non-ST-segment elevation myocardial infarction, and unstable angina.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Total MACE at 2 years | 1 month,1year,2 years
  The total MACE (Major Adverse Cardiovascular Events) at 2 years post-surgery, including both culprit lesions and non-culprit lesions, is defined as a composite endpoint consisting of death, non-fatal myocardial infarction, and unplanned revascularization.

SECONDARY OUTCOMES:
CL-MACE at 2 years post-PCI; NCL-MACE at 2 years post-PCI | 1 month,1year,2 years
  The CL-MACE at 2 years post-PCI and NCL-MACE at 2 years post-PCI， including both culprit lesions and non-culprit lesions, is defined as a composite endpoint consisting of death, non-fatal myocardial infarction, and unplanned revascularization.
Major Adverse Cardiovascular Events | 1 month,1year,2 years,5 years
  MACE includes recurrent angina, acute myocardial infarction, severe arrhythmias, heart failure, coronary death, and so on.
Death | 1 month,1year,2 years,5 years
  Death includes all-cause mortality, cardiovascular mortality, non-cardiovascular mortality, and deaths of unknown causes.
Non-fatal Myocardial Infarction | 1 month,1year,2 years,5 years
  Non-fatal Myocardial Infarction (NBMI) refers to an event where the heart muscle suffers severe ischemia and necrosis due to the acute occlusion of the coronary artery, but does not result in the patient's death. This type of heart attack is usually accompanied by changes on the electrocardiogram (ECG) and elevated cardiac biomarkers (such as troponin), but without significant elevation of the ST segment, which distinguishes it from ST-segment elevation myocardial infarction (STEMI).
Unplanned Revascularization | 1 month,1year,2 years,5 years
  Unplanned revascularization is defined as revascularization performed outside the scope of the initial standard treatment for PCI, or staged revascularization that occurs more than 60 days (or the number of days planned by the surgeon) after the first PCI. Unplanned revascularization refers to PCI or CABG driven by persistent ischemic symptoms.
Any Revascularization | 1 month,1year,2 years,5 years
  Any revascularization includes planned revascularization, unplanned revascularization, target lesion revascularization, ischemia-driven target lesion revascularization, and clinically driven target lesion revascularization.
Stent Thrombosis As Defined by ARC-2 | 1 month,1year,2 years,5 years
  Stent thrombosis is classified by the time of occurrence into acute thrombosis (occurring within 24 hours after PCI), subacute thrombosis (occurring between 1-30 days after PCI), late thrombosis (occurring between 31 days and 365 days after PCI), or very late thrombosis (occurring more than 365 days after PCI).

CONTACTS AND LOCATIONS:
Overall Officials: Yun Dai Chen, MD, PHD, Study Chair — People's Liberation Army General Hospital; Yong Zeng, PD, Principal Investigator — Beijing Anzhen Hospital; Lei Song, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Jun Jiang, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Yuquan He, MD, Principal Investigator — China-Japan Union Hospital, Jilin University; Wei Liu, MD, Principal Investigator — Beijing Jishuitan Hospital; Da Yin, MD, Principal Investigator — Shenzhen People's Hospital; Yining Yang, MD, Principal Investigator — People's Hospital of Xinjiang Uygur Autonomous Region; Jie Deng, MD, Principal Investigator — Xi'an Jiaotong University Second Affiliated Hospital; Ning Yang, MD, Principal Investigator — Tianjin Chest Hospital; Hua Yan, Principal Investigator — Wuhan Asian Heart Hospital
Locations (11):
- China (11):
  - Shenzhen People's Hospital, Shenzhen, Guandong
  - Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Asian Heart Hospital, Wuhan, Hubei
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Xi'an Jiaotong University Second Affiliated Hospital, Xi'an, Shaanxi
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang Uygur Autonomous Region
  - The Second Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Jishuitan Hospital, Beijing
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing
  - People's Liberation Army General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mol JQ, Volleberg RHJA, Belkacemi A, Hermanides RS, Meuwissen M, Protopopov AV, Laanmets P, Krestyaninov OV, Dennert R, Oemrawsingh RM, van Kuijk JP, Arkenbout K, van der Heijden DJ, Rasoul S, Lipsic E, Rodwell L, Camaro C, Damman P, Roleder T, Kedhi E, van Leeuwen MAH, van Geuns RM, van Royen N. Fractional Flow Reserve-Negative High-Risk Plaques and Clinical Outcomes After Myocardial Infarction. JAMA Cardiol. 2023 Nov 1;8(11):1013-1021. doi: 10.1001/jamacardio.2023.2910. PMID 37703036
- [Result] Erlinge D, Maehara A, Ben-Yehuda O, Botker HE, Maeng M, Kjoller-Hansen L, Engstrom T, Matsumura M, Crowley A, Dressler O, Mintz GS, Frobert O, Persson J, Wiseth R, Larsen AI, Okkels Jensen L, Nordrehaug JE, Bleie O, Omerovic E, Held C, James SK, Ali ZA, Muller JE, Stone GW; PROSPECT II Investigators. Identification of vulnerable plaques and patients by intracoronary near-infrared spectroscopy and ultrasound (PROSPECT II): a prospective natural history study. Lancet. 2021 Mar 13;397(10278):985-995. doi: 10.1016/S0140-6736(21)00249-X. PMID 33714389
- [Result] Mol JQ, Belkacemi A, Volleberg RH, Meuwissen M, Protopopov AV, Laanmets P, Krestyaninov OV, Dennert R, Oemrawsingh RM, van Kuijk JP, Arkenbout K, van der Heijden DJ, Rasoul S, Lipsic E, Teerenstra S, Camaro C, Damman P, van Leeuwen MA, van Geuns RJ, van Royen N. Identification of anatomic risk factors for acute coronary events by optical coherence tomography in patients with myocardial infarction and residual nonflow limiting lesions: rationale and design of the PECTUS-obs study. BMJ Open. 2021 Jul 7;11(7):e048994. doi: 10.1136/bmjopen-2021-048994. PMID 34233996
- [Result] Aguirre AD, Arbab-Zadeh A, Soeda T, Fuster V, Jang IK. Optical Coherence Tomography of Plaque Vulnerability and Rupture: JACC Focus Seminar Part 1/3. J Am Coll Cardiol. 2021 Sep 21;78(12):1257-1265. doi: 10.1016/j.jacc.2021.06.050. PMID 34531027